CLINICAL TRIAL: NCT04546906
Title: Safety and Efficacy Study of CD22 CAR-T Cells for Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD22 CAR-T for B-ALL
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: B-ALL
Keywords: CD22 CAR-T， B-ALL

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD22 CAR-T (Experimental): Patients will be treated with CD22 CAR-T cells
  Interventions: Biological: CD22 CAR-T

INTERVENTIONS:
Biological: CD22 CAR-T — Biological: CD22 CAR-T; Drug: Cyclophosphamide,Fludarabine; Procedure: Leukapheresis

SUMMARY:
This is an open, single-arm, clinical study to evaluate efficacy and safety of anti CD22 CAR-T cell in the treatment of recurrent or refractory B-ALL

DETAILED DESCRIPTION:
The CARs consist of an anti-CD22 single-chain variable fragment（scFv）, a portion of the human CD137（4-1BB） molecule, and the intracellular component of the human CD3ζ molecule. Prior to CAR-T cell infusion, the patients will be subjected to preconditioning treatment. After CAR-T cell infusion, the patients will be evaluated for adverse reactions and efficacy.

The Main research objectives:

To evaluate the safety and efficacy of CD22CAR-T in patients with recurrent or refractory B-ALL

The Secondary research objectives:

To investigate the cytokinetic characteristics of CD22CAR-T in patients with recurrent or refractory B-ALL

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed and refractory acute B-lymphoblastic leukemia who have any of the following:

   1. B-ALL patients with relapse (including bone marrow morphological relapse 1 and minimal residual relapse 2) after remission by chemotherapy or autologous stem cell transplantation;
   2. Primary B-ALL patients who can not be completely relieved by more than two times of repeated chemotherapy;
   3. High risk primary B-ALL patients who have not been relieved but are not suitable for re intensive therapy after 1-2 times of chemotherapy;
2. Flow cytometry (FCM) showed CD 22 positive in bone marrow or peripheral blood;
3. There should be at least one assessable lesion in B-ALL patients with simple extramedullary recurrence;
4. The activity state score of the Eastern Cooperative Oncology Group (ECOG) was less than or equal to 2;
5. The estimated survival time is more than 3 months;
6. Need to sign informed consent.

Exclusion Criteria:

1. Serious cardiac insufficiency；
2. Has a history of severe pulmonary function damaging;
3. Other malignant tumors;
4. Serious infection or persistent infection and can not be effectively controlled；
5. Merging severe autoimmune diseases or immunodeficiency disease;
6. Patients with active hepatitis (HBV DNA or HCV RNA positive);
7. Patients with HIV infection or syphilis infection;
8. Has a history of serious allergies on Biological products (including antibiotics);
9. Being pregnant and lactating or having pregnancy within 12 months;
10. Any situations that the researchers believe will increase the risks for the subject or affect the results of the study（including a history of serious mental illness, substance abuse and addiction）

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First month post CAR-T cells infusion
  To evaluate the possible adverse events occurred within first one month after CD22 CAR-T infusion, including the incidence and severity of symptoms such as cytokine release syndrome and neurotoxicity
Efficacy: Remission Rate | 3 months post CAR-T cells infusion
  Remission Rate including complete remission(CR)、CR with incomplete blood count recovery(CRi)、No remission(NR)

SECONDARY OUTCOMES:
Efficacy:duration of response (DOR) | 24 months post CAR-T cells infusion
  duration of response (DOR)
Efficacy: progression-free survival (PFS) | 24 months post CAR-T cells infusion
  progression-free survival (PFS) time
CAR-T proliferation | 3 months post CAR-T cells infusion
  the copy number of CD19 CAR- T cells in the genomes of PBMC by qPCR method and percentage of CD19 CAR- T cells measured by flow cytometry method
Cytokine release | First month post CAR-T cells infusion
  Cytokine( IL-6,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by flow cytometry method

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, PhD&MD, Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (2):
- China (2):
  - Hebei yanda Ludaopei Hospital, Heibei, Sanhe
  - BeiJing Ludaopei Hospital, Beijing, Yizhuang